CLINICAL TRIAL: NCT07150767
Title: A Clinical Study to Explore the Safety, Tolerability, and Efficacy of Recombinant Human nsIL12 Oncolytic Adenovirus Injection (BioTTT001) Combined With Neoadjuvant Treatment for Locally Advanced Breast Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The applicant voluntarily withdrew the case
Sponsor: Beijing Bio-Targeting Therapeutics Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-01-108
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Breast Cancer (LABC)
Keywords: Recombinant Human nsIL12 Oncolytic Adenovirus Injection (BioTTT001)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BioTTT001 is administered as a single Intratumoral injection. (Experimental): HER-2 positive breast cancer group、triple-negative breast cancer group、Hormone receptor-positive breast cancer group: BioTTT001: According to the dose escalation requirements, a total of three injections of BioTTT001 d1, d3, and d5 in the first cycle, and the sequential neoadjuvant regimen was started on d22 days. Subsequently, according to the administration time of the neoadjuvant regimen, one dose of the same dose of BioTTT001 was supplemented every cycle d15.HER-2 positive breast cancer group：THP regimen: albumin paclitaxel 125 mg/m2, d1, d8;Trastuzumab 8mg/kg for the first dose, then 6 mg/kg, d1;Pertuzumab is 840mg for the first dose, followed by 420mg, d1, Q3w.4 cycles in total.triple-negative breast cancer group：albumin paclitaxel 125 mg/m2,d1,d8;Carboplatin AUC=5 d1;Toripalimab 240mg, d1, Q3w, a total of 4 cycles.Hormone receptor-positive breast cancer group:
  Docetaxel 75mg/m2, d1;Doxorubicin 50mg/m2,d1;Cyclophosphamide 500mg/m2, d1, Q3w, a total of 6 cycles.
  Interventions: Biological: BioTTT001 injection

INTERVENTIONS:
Biological: BioTTT001 injection — BioTTT001 is administered as a multiple Intratumoral injection. The dose groups to be infusion were 5.0×10^10 viral particle (VP) ,2.0×10^11 VP and 5×10^11 VP based on the 3+3 dose escalation principle.

SUMMARY:
A clinical study to explore the safety, tolerability, and efficacy of recombinant human nsIL12 oncolytic adenovirus injection (BioTTT001) combined with neoadjuvant treatment for locally advanced breast cancer.This study is a single-arm, open-label, single-center dose-escalation and expansion trial.

DETAILED DESCRIPTION:
Three study drug dose groups were preset, namely 5×10^10VP、2×10^11VP and 5×10^11VP and the "3+ 3" dose escalation method was adopted according to the principle of dose escalation and the sequential principle from low to high.In order to protect the safety of subjects, in theory, in order to protect the safety of subjects, the second subject can be enrolled at least 2 weeks after the administration of the first subject in each dose group at least 2 weeks after administration in the DLT observation phase of the same dose group. The DLT observation period for each subject is 21 days after the first dose, and the next dose escalation can only be entered after the last subject in each dose group completes the DLT observation period. At least 3 subjects were enrolled in each dose group, and each subject received only one corresponding dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age> 18 years old (including cut-off value), female;
2. Patients with resectable stage II.a-III.c primary non-metastatic breast cancer confirmed by histopathology and/or cytology (clinical stage: cT2-T4, cN0-N3, M0);
3. At least one evaluable lesion according to RECIST 1.1 in solid tumors
4. There are lesions suitable for intratumoral injection as assessed by the investigator (the evaluable lesion and the intratumoral injection lesion can be the same lesion);
5. ECOG PS score 0-1 points;
6. The values of the laboratory tests performed for screening must meet the following standards:

   Routine blood tests:

   WBC≥3.0×10^9/L； ANC ≥ 1.5×10^9/L, and no cytokine correction therapy within 1 week prior to screening; Subjects with Hb≥90g/L and no blood transfusion within 1 week; Subjects who have a white > of 80g/L before blood transfusion and have received blood transfusion within 3 days before screening to meet the standard (Hb≥90g/L); PLT≥90×10^9/L and no platelet transfusion or thrombopoietin corrective therapy within 1 week prior to screening.

   Blood biochemical tests:

   ALT and AST≤ 3×ULN (or ≤5×ULN if with liver metastases); Serum creatinine ≤1.5×ULN or CCr>50mL/min; TBIL≤1.5×ULN； APTT≤1.5×ULN, while INR or PT≤1.5×ULN;
7. Expected survival ≥ 3 months;
8. All subjects and their partners have no birth plan from screening to the end of the trial and agree to take effective non-drug contraceptive measures (such as condoms, intrauterine devices without medication, etc.) during the trial, except for those who have taken permanent contraceptive measures, such as bilateral tubal ligation, vasectomy, etc.;
9. Volunteer to participate in clinical research and sign the informed consent form.

Exclusion Criteria:

1. Known allergy to the study drug or its components;
2. Those who have received other adenovirus drugs;
3. Patients with active or previously suffered autoimmune diseases that may recur (such as systemic lupus erythematosus, rheumatoid arthritis, etc.), except for type 1 diabetes, hypothyroidism that only needs to be treated with hormone replacement, skin diseases that do not require systemic treatment (such as vitiligo, psoriasis, or alopecia);
4. Treatment with nitrosoureas or mitomycin C within 6 weeks prior to starting study treatment; Received oral fluorouracil and small molecule targeted drug therapy within 2 weeks or 5 half-lives of the drug (whichever is longer) prior to starting study treatment; Received traditional Chinese medicine treatment with anti-tumor indications within 2 weeks before starting study treatment; Received anti-tumor therapy such as chemotherapy, radiotherapy, biological therapy, endocrine therapy, etc. other than the above-mentioned drugs within 28 days before starting study treatment, or received any other unmarketed investigational drugs;
5. Those who have not recovered from the adverse reactions of previous treatment (treatment-related toxicity grade ≤ grade 2, except for alopecia, pigmentation and other tolerable events as judged by the investigator or laboratory abnormalities allowed according to the protocol);
6. Other malignant tumors occurred within 5 years before enrollment, except for carcinoma in situ of the cervix that has been effectively resected and does not require continued anti-tumor treatment, low-risk to very low-risk gastrointestinal stromal tumors (primary tumors at any site, tumor size is ≤5cm, and the number of nuclear division images per 50 high-power field ≤5), in situ or early (stage I) breast cancer, basal cell carcinoma of the skin, papillary thyroid carcinoma;
7. Those who have undergone any major surgery (except for needle biopsy, etc.) or severe trauma within 4 weeks before the first dose;
8. Patients who have been treated with high-dose systemic corticosteroids (prednisone> 10mg/day or equivalent dose of similar drugs) or other immunosuppressants within 2 weeks before the first dose. In addition to the following conditions: treatment with topical, ocular, intraarticular, intranasal and inhaled corticosteroids; short-term use of corticosteroids for prophylactic treatment, such as the use of contrast agents;
9. Congestive heart failure with cardiac function ≥ NYHA class III; Acute myocardial infarction or unstable angina within 6 months prior to dosing; Left ventricular ejection fraction (LVEF) <50%; Corrected QTc interval (corrected by Fridericia's formula) > 450 msec for males and >470 msec for females, or risk factors for torsades de pointes, such as clinically significant hypokalemia, family history of long QT syndrome, or familial history of cardiac arrhythmias (eg, preexcitation syndrome) as judged by the investigator;
10. Active tuberculosis, drug-induced interstitial lung disease;
11. Presence of active inflammatory bowel disease (such as Crohn's disease or ulcerative colitis);
12. Active infection requiring systemic anti-infective therapy; Unexplained fever > 38.5°C (neoplastic fever subjects are judged by the investigator to be included in the study);
13. Immunosuppressed, such as severe combined immunodeficiency disease or concurrent opportunistic infections;
14. Active hepatitis B (positive for HBsAg and 100IU/mL for HBV DNA titer test ≥100IU/mL) and/or positive for anti-HCV (and positive for HCV RNA) at screening; Patients with active syphilis infection or positive human immunodeficiency virus (HIV) screening results;
15. Pleural effusion and ascites with clinical symptoms that require repeated drainage;
16. Central nervous system metastases or meningeal metastases with clinical symptoms, or other evidence of central nervous system metastases or meningeal metastases with clinical symptoms, or other evidence that the patient's central nervous system metastases or meningeal metastases have not been controlled, and are judged by the investigator to be unsuitable for enrollment;
17. Pregnant or lactating women;
18. Patients with previous organ transplantation;
19. The investigator believes that the patient is not suitable for this trial for any reason.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03-26 (Actual); Primary Completion 2027-03-26 (Estimated); Study Completion 2027-03-26 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | The DLT observation period for each subject is 21 days after the first dose
  Incidence and severity of dose-limiting toxicities (DLTs) and various adverse events assessed based on NCI-CTCAE V5.0.Maximum tolerated dose (MTD) and recommended dose (RP2D).

CONTACTS AND LOCATIONS:
Locations (1):
- The Second People's Hospital of Shandong Province, Jinan, Shandong, China